CLINICAL TRIAL: NCT03342196
Title: A Phase II Study of Thiotepa Added to Fludarabine and Melphalan as the Preparative Regime for Alternative Donor Transplantation
Brief Title: Thiotepa Plus Fludarabine+ Melphalan as the Preparative Regime for Alternative Donor Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE10Z17
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Leukemia
Keywords: Thiotepa; Fludarabine; Melphalan
MeSH Terms: conditions — Leukemia | interventions — Melphalan; Thiotepa; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thiotepa + Fludarabine + Melphalan (Experimental): Melphalan 100 mg/m2 on day -8 Thiotepa 10 mg/kg on day -7 Fludarabine 160 mg/m2 in divided doses given on days -6, -5, -4 and -3.
  Interventions: Drug: Melphalan; Drug: Thiotepa; Drug: Fludarabine

INTERVENTIONS:
Drug: Melphalan — Alkylating agent which is a derivative of mechlorethamine that inhibits DNA and RNA synthesis via formation of carbonium ions; cross-links strands of DNA; acts on both resting and rapidly dividing tumor cells.
  Melphalan may cause a lowering of the white blood cell or platelet counts, leading to an increased risk of infection and frequent bruising or bleeding. It may cause damage to the GI tract causing mouth sores, nausea, vomiting, and diarrhea. Other side effects may include loss of appetite, liver abnormalities, hair loss, swelling, fatigue, sleepiness, skin rash.
  Other Names: Alkeran; Evomela
Drug: Thiotepa — Thiotepa is an alkylating agent which produces cross-linking of DNA strands leading to inhibition of DNA, RNA, and protein synthesis; thiotepa is cell-cycle independent.
  Thiotepa may cause a lowering of the white blood cell or platelet counts, leading to an increased risk of infection and frequent bruising or bleeding. It may cause damage to the GI tract causing mouth sores, nausea, vomiting, and diarrhea. Other side effects may include loss of appetite, liver abnormalities, hair loss, swelling, fatigue, sleepiness, skin rash.
  Other Names: Tepadina
Drug: Fludarabine — Fludarabine is an antineoplastic fluorinated nucleoside analog and inhibits DNA synthesis through inhibition of polymoerase alpha after incorporation into DNA.
  Fludarabine may cause a lowering of the white blood cell or platelet counts, leading to an increased risk of infection and frequent bruising or bleeding. Other side effects may include loss of appetite, liver abnormalities, hair loss, swelling, fatigue, sleepiness, skin rash, and lower limb weakness.
  Other Names: Fludara

SUMMARY:
In the United States, thiotepa has been utilized in reduced intensity conditioning regimens for alternative donor courses (double umbilical cord blood transplant (dUCBT) and haplo-identical transplants).

The hypothesis is that thiotepa at a dose of 10mg/kg, in combination with melphalan (100mg/m2) and fludarabine (160mg/m2) as a reduced intensity conditioning regimen for alternative donor transplant is safe and effective in patients with hematologic malignancies.

Given that this regimen has been investigated extensively, and the current study proposes to confirm those previous observations with a small modification (melphalan dose reduction due to previous mucositis rates with higher doses), this will be a phase II study designed to measure disease-free-survival.

DETAILED DESCRIPTION:
Primary Objective:

To assess the effectiveness of Thiotepa, Fludarabine, and Melphalan in alternative donor transplants as measured by leukemia free survival.

Secondary Objective:

To assess the 1- year OS, Relapse, TRM, aGVHD and cGVHD rates and the rates of neutrophil and platelet engraftment.

Study Design This is a Phase II study of Thiotepa, Fludarabine, and Melphalan in alternative donor transplants.

Subjects will be assessed for safety and tolerability (including adverse events, serious adverse events, and clinical/laboratory assessments) using a continuous monitoring approach. Subjects will be followed for up to 1 year or until progression of disease, relapse, or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following hematologic malignancies:

  * Acute myelogenous leukemia (AML): High-risk AML including:

    * Antecedent hematological disease (e.g., myelodysplasia (MDS))
    * Treatment-related leukemia
    * Complete Remission (CR1) with poor-risk cytogenetics or molecular markers (e.g. Flt 3 mutation, 11q23, del 5, del 7, complex cytogenetics)
    * Second complete remission (CR2) or third complete remission (CR3)
    * Induction failure or 1st relapse with ≤ 10% blasts in the marrow
  * Acute lymphoblastic leukemia (ALL)

    * High-risk CR1 including:

      * Poor-risk cytogenetics (e.g., Philadelphia chromosome t(9;22)or 11q23 rearrangements)
      * Presence of minimal disease by flow cytometry after 2 or more cycles of chemotherapy
    * No CR within 4 weeks of initial treatment
    * Induction failure with ≤ 10% blasts in the marrow
    * CR2 or CR3
  * Myelodysplastic syndromes (MDS), Intermediate, High or Very High Risk by the revised international prognostic scoring system (IPSS-R)
  * Mixed Phenotypic Leukemia / Biphenotypic Leukemiain CR
  * Chronic Myelogenous Leukemia (CML) in second chronic phase after accelerated or blast crisis.
  * Myelofibrosis (MF):

    * Intermediate-1, Intermediate-2 or high risk by Dynamic International Prognostic Scoring System (DIPSS-plus) or
    * Monosomal karyotype or
    * Presence of inv(3)/i(17q) abnormalities or
    * Other unfavorable karyotype OR leukocytes ≥40 × 10(9) /L and
    * Circulating blasts ≤ 9%
  * Chronic Myelomonocytic Leukemia
  * Relapsed or Refractory Lymphoid Malignancies (including non-Hodgkin Lymphoma, Hodgkin Lymphoma and Chronic Lymphocytic Leukemia) meeting the following criteria:

    * Disease status: Stable Disease, Partial Remission or 2nd and 3rd Complete Remission. OR
    * Have relapsed after autologous transplant or who have failed to collect for an autologous transplant.
* Age > 1 years, < 65yrs
* KPS Performance status ≥80
* Patients without a matched related or unrelated donor
* Patient with either one or both:

  * Two 5/8 human leukocyte antigen (HLA) high resolution matched umbilical cord blood (UCB) grafts with a cell dose of 2.0x10^7 total number of nucleated cells per kilogram (TNC/kg) each, or
  * A related haplo-identical donor
* Concurrent Therapy for Extramedullary Leukemia or central nervous system (CNS) Lymphoma: Concurrent therapy or prophylaxis for testicular leukemia, CNS leukemia, and CNS lymphoma including standard intrathecal chemotherapy and/or radiation therapy will be allowed as clinically indicated. Such treatment may continue until the planned course is completed. Subjects must be in CNS remission at the time of protocol enrollment if there is a history of CNS involvement. Maintenance therapy after transplant is allowed.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with inadequate Organ Function as defined by:

  * Creatinine clearance <50ml/min
  * Bilirubin > twice institutional upper limit of normal
  * aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) ≥ three times institutional upper limit of normal
  * Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) ≥ three times institutional upper limit of normal
  * Pulmonary function: diffusing capacity of the lung for carbon monoxide corrected for hemoglobin (DLCOc) < 60% normal
  * Cardiac: left ventricular ejection fraction < 50%
  * Karnofsky Performance Statue (KPS) < 80
* Patients with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because chemotherapy involved with Reduced Intensity Conditioning (RIC) have the significant potential for teratogenic or abortifacient effects.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds
* Presence of donor-specific antibodies against chosen graft source.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Thiotepa + Fludarabine + Melphalan: Melphalan 100 mg/m2 on day -8 Thiotepa 10 mg/kg on day -7 Fludarabine 160 mg/m2 in divided doses given on days -6, -5, -4 and -3.
  Melphalan: Alkylating agent which is a derivative of mechlorethamine that inhibits DNA and RNA synthesis via formation of carbonium ions; cross-links strands of DNA; acts on both resting and rapidly dividing tumor cells.
  Melphalan may cause a lowering of the white blood cell or platelet counts, leading to an increased risk of infection and frequent bruising or bleeding. It may cause damage to the GI tract causing mouth sores, nausea, vomiting, and diarrhea. Other side effects may include loss of appetite, liver abnormalities, hair loss, swelling, fatigue, sleepiness, skin rash.
  Thiotepa: Thiotepa is an alkylating agent which produces cross-linking of DNA strands leading to inhibition of DNA, RNA, and protein synthesis; thiotepa is cell-cycle independent.
  Thiotepa may cause a lowering of the white blood cell or platelet counts, leading to an increased risk of infection and frequent bruising or bleeding. It may cause damage to the GI tract causing mouth sores, nausea, vomiting, and diarrhea. Other side effects may include loss of appetite, liver abnormalities, hair loss, swelling, fatigue, sleepiness, skin rash.
  Fludarabine: Fludarabine is an antineoplastic fluorinated nucleoside analog and inhibits DNA synthesis through inhibition of polymoerase alpha after incorporation into DNA.
Period: Overall Study
Arm/Group | Thiotepa + Fludarabine + Melphalan
Started | 40
Completed | 39
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  10-19 | 1
  20-29 | 4
  30-39 | 7
  40-49 | 3
  50-59 | 12
  60-69 | 12
  70-79 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Disease Free Survival
Description: Leukemia Free Survival (LFS) at 1 year is the percentage of patients alive and without evidence of hematologic malignancy at 1 year after transplant.
Time Frame: Up to 1 year after transplant
Population: 1 participant was non evaluable for this measure
Measure: Number; unit: percentage of paticipants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 38
percentage of paticipants | 65.8

2. Primary Outcome: Percentage of Patients With Leukemia Free Survival
Time Frame: Up to 1 year after transplant
Population: Trial changes eligibility amended to include other hematological diseases - of the 40 pts on study - 39 went to treatment, 1 on treatment non evaluable, and only 29 had Leukemia (ALL/CML/CMML and AML)
Measure: Number; unit: percentage of paticipants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 29
percentage of paticipants | 65.5

3. Secondary Outcome: Average Overall Survival
Description: Overall Survival (OS) at 1 year is the percentage of patients alive at 1 year after transplant.
Time Frame: Up to 1 year after transplant
Population: 1 participant was non evaluable for this measure
Measure: Number; unit: percentage of participants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 38
percentage of participants | 73.7

4. Secondary Outcome: Relapse Incidence
Description: Relapse incidence at 1 year is the percentage of patients who experience relapse of their hematologic malignancy up to 1 year after transplant.
Time Frame: Up to 1 year after transplant
Population: 9 participants were non evaluable for this measure
Measure: Number; unit: percentage of participants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 30
percentage of participants | 13.16

5. Secondary Outcome: Treatment Related Mortality
Description: Treatment Related Mortality (TRM) at 1 year is the percentage of patients who expire from treatment related toxicity attributed to transplant up to 1 year after transplant.
Time Frame: Up to 1 year after transplant
Population: 1 participant was non evaluable for this measure
Measure: Number; unit: percentage of paticipants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 38
percentage of paticipants | 21.05

6. Secondary Outcome: Incidence of Acute GVHD
Description: Acute graft versus host disease (aGVHD) 1 year cumulative incidence is the percentage of patients who experience any aGVHD up to 1 year after transplant.
Time Frame: Up to 1 year after transplant
Population: 1 participant was non evaluable for this measure
Measure: Number; unit: percentage of participants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 38
percentage of participants | 76.31

7. Secondary Outcome: Incidence of Chronic GVHD
Description: Chronic graft versus host disease (cGVHD) 1-year cumulative incidence is the percentage of patients who experience any cGVHD up to 1 year after transplant.
Time Frame: Up to 1 year after transplant
Population: 1 participant was non evaluable for this measure
Measure: Number; unit: percentage of participants
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 38
percentage of participants | 21.05

8. Secondary Outcome: Rate of Neutrophil Engraftment
Description: Neutrophil engraftment will be calculated as the days from transplant where the absolute neutrophil count (ANC) reaches >500cells/ul x 3 days.
Time Frame: Up to 1 year after transplant
Population: 4 participants were non evaluable for this measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 35
Days | 20.6 (5.69)

9. Secondary Outcome: Rate of Platelet Engraftment
Description: Platelet engraftment will be calculated as the days from transplant where the platelet count reaches 20,000 platelets /ul without the need of transfusion of platelets for 7 days.
Time Frame: Up to 1 year after transplant
Population: 5 participants were non evaluable for this measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Thiotepa + Fludarabine + Melphalan
Number analyzed (Participants) | 34
Days | 42.32 (31.4)

ADVERSE EVENTS:
Time Frame: Participants were followed for this study for 1 year following the allogeneic transplant, relapse, or death, whichever occured first.
Arm/Group | Thiotepa + Fludarabine + Melphalan
All-Cause Mortality (participants affected / at risk) | 14/40
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thiotepa + Fludarabine + Melphalan (N=40)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (2)
Encephalitis infection (Infections and infestations) | 1 (3)
Enterocolitis infectious (Infections and infestations) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Heart failure (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Immune system disorders - Other, specify (Immune system disorders) | 1 (4) — GVHD
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Adenovirus Colitis
Enterocolitis infectious (Infections and infestations) | 1 (1) — D. difficile infection - IV antibiotic
Enterocolitis infectious (Infections and infestations) | 1 (2) — Yersinia Entercolitica Infection
Fungemia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Stenotrophomonas Maltophilia
Lung infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (10)
Multi-organ failure (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6)
Pericardial effusion (Cardiac disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) — Epilepsy associated infection, currently inconclusive on what infection caused the status epilepticus.
Sepsis (Infections and infestations) | 1 (2) — Septic shock due to Stenotrophomonas maltophilia.
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (3)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (2)
Syncope (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thiotepa + Fludarabine + Melphalan (N=40)
Abdominal pain (Gastrointestinal disorders) | 6 (10)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (9)
Alanine aminotransferase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Anxiety (Psychiatric disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bacteremia (Infections and infestations) | 1 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3)
Confusion (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Investigations) | 4 (4)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (17)
Dizziness (Nervous system disorders) | 2 (2)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema limbs (General disorders) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye infection (Eye disorders) | 1 (1)
Fatigue (General disorders) | 6 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 10 (17)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fungemia (Infections and infestations) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (16)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Immune system disorders - Other, specify (Immune system disorders) | 3 (6)
Infections and infestations - Other, specify (Infections and infestations) | 4 (6)
Investigations - Other, specify (Investigations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 5 (9)
Multi-organ failure (General disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (3)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (3)
Serum amylase increased (Investigations) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 3 (5)
Sudden death NOS (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 3 (3)
Thrush (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Viremia (Infections and infestations) | 1 (5)
Vomiting (Gastrointestinal disorders) | 6 (7)
Weight loss (Investigations) | 4 (5)
White blood cell decreased (Investigations) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03342196/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03342196/ICF_001.pdf